CLINICAL TRIAL: NCT01764165
Title: Pathogenesis and Outcomes of Sleep Disordered Breathing in COPD
Brief Title: Pathogenesis and Outcomes of Sleep Disordered Breathing in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Hartmut Schneider, Assistant Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HL105546-01 (NIH); NA_00040333 (Other: Johns Hopkins Medicine-IRB 5)
Record Dates: First submitted 2010-07-16; First posted 2013-01-09 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: COPD
Keywords: COPD; Sleep; Supplemental oxygen; Breathing mechanics; nasal insufflation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Oxygen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oxygen (Active Comparator): nocturnal oxygen of 2 L/min
  Interventions: Other: Oxygen
- High Flow of room air (Experimental): Warm and humidified air at a rate of 20 L/min through a small nasal cannula (similar to oxygen cannula)
  Interventions: Other: High flow of room air

INTERVENTIONS:
Other: Oxygen — oxygen at a rate of 2 L/min will be delivered through a small nasal cannula throughout sleep.
  Other Names: supplemental oxygen; nocturnal oxygen
  Arms: oxygen
Other: High flow of room air — Warm and humidified air at rates of 20 L/min will be delivered through a small nasal cannula throughout sleep
  Other Names: TNI: Transnasal insufflation; Open CPAP; Optiflow
  Arms: High Flow of room air

SUMMARY:
This research is being conducted to examine the effects of nasal insufflation of warm and humidified air through a small nasal cannula on sleep, breathing pulmonary function, and daytime exercise capability.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is associated with significant morbidity including substantial daytime fatigue exertional intolerance and ventilatory impairment, which hits a nadir in the morning. Nocturnal disturbances in sleep and breathing are common in COPD, although the impact of these disturbances on COPD morbidity remains largely unknown. The hypothesis is that COPD induces specific sleep and breathing disturbances that remain a substantial source of morbidity in this disorder.

Current therapy for treating nocturnal disturbances in sleep and breathing in COPD including nocturnal oxygen has failed to improve morning fatigue and pulmonary function. This study promises to significantly alter our approach to the diagnosis and management of sleep disordered breathing in COPD.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adults over the age of 21
* BMI < 40 kg/m2

Exclusion Criteria:

* Diagnosed with sleep apnea (apnea and hypopneas of >10 events/hr).
* A sleep efficiency of <30%, or a prior diagnosis of disorders that impair sleep architecture.
* Unstable cardiovascular disease (decompensated heart failure, myocardial infarction within the past 3 months, revascularization procedure within the past 3 months, unstable arrhythmias, uncontrolled hypertension (BP > 190/110)).
* Severe renal insufficiency requiring dialysis.
* Liver cirrhosis.
* A recent acute illness in a 6 weeks period prior to the sleep studies.
* We will exclude subjects with severe daytime hypoxemia (Oxyhemoglobin saturation (SaO2) <80% or partial pressure of oxygen (PaO2) <55 mmHg at rest).
* Chronic use of sedatives or respiratory depressants that would affect sleep quality (e.g., benzodiazepines or other hypnotics or narcotics).
* Pregnancy.
* Tracheostomy or other significant oropharyngeal or nasopharyngeal surgery, in the last 6 months.
* Narcolepsy and other neurological disorders such as Parkinson's Disease.
* Severe hepatic insufficiency.
* Bleeding disorders or Coumadin use.
* Allergy to lidocaine or benzocaine.
* Language/dementia/psychiatric issues - the participant must be able to provide consent.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The evening to morning differences in expiratory airflow obstruction (FEV1/FVC) | 4 years
  Lung function declines over the course of the night. We hypothesize that delivering warm and humidified air at a rate of 20 L/min over the entire night improves morning FEV1 compared to oxygen.

SECONDARY OUTCOMES:
The percent rate of inspiratory flow limitation. | 4 Years
  Patients with COPD often exhibit inspiratory air flow limitation during sleep. We hypothesize that delivering warm and humidified air at a rate of 20 L/min reduces the degree of inspiratory air flow limitation compared to oxygen.
Effect of High flow nasal insufflation of air on exercise capacity (6 minute walk test). | One Year
  Patients with COPD have impaired exercise tolerance in the morning. We hypothesize that delivering warm and humidified air at a rate of 20 L/min over the entire night extends morning 6 minute walk length.

OTHER OUTCOMES:
Sleep efficiency | 4 years
  We hypothesize that delivering warm and humidified air at a rate of 20 L/min over the entire night improves sleep efficiency compared to oxygen treatment.
Episodes of dynamic hyperinflation | 4 years
  The combination of in- and expiratory flow limitation can lead to dynamic hyperinflation during sleep. We hypothesize that compared to oxygen, high flow nasal insufflation of warm and humidified air at a rate of 20 L/min will reduce the number of breaths associated with dynamic hyperinflation.

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Schneider, M.D., Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Background] Schneider H, Krishnan V, Pichard LE, Patil SP, Smith PL, Schwartz AR. Inspiratory duty cycle responses to flow limitation predict nocturnal hypoventilation. Eur Respir J. 2009 May;33(5):1068-76. doi: 10.1183/09031936.00063008. Epub 2009 Jan 7. PMID 19129290